CLINICAL TRIAL: NCT03906695
Title: A Multicenter, Open-label, Dose-escalation, Phase 1 Trial to Investigate the Tolerability and Safety of ASTX727 in Subjects With Lower-risk Myelodysplastic Syndromes
Brief Title: Phase 1 Trial of ASTX727 in Subjects With Lower-risk Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 393-102-00002; JapicCTI-194654 (Other: Japic)
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Lower-risk Myelodysplastic
MeSH Terms: interventions — decitabine and cedazuridine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 10-Day Schedule (Experimental): 10-Day Schedule
  Investigational Medicinal Products (IMP) will be administered for 10 days in total per 4 weeks, i.e. a 28-day cycle.
  Interventions: Drug: ASTX727
- 5-Day Schedule A (Experimental): 5-Day Schedule A
  IMP will be administered for 5 days in total per 4 weeks, i.e. a 28-day cycle.
  Interventions: Drug: ASTX727
- 5-Day Schedule B (Experimental): 5-Day Schedule B
  IMP will be administered for 5 days in total per 4 weeks, i.e. a 28-day cycle.
  Interventions: Drug: ASTX727
- 5-Day Schedule C (Experimental): 5-Day Schedule C
  IMP will be administered for 5 days in total per 4 weeks, i.e. a 28-day cycle.
  Interventions: Drug: ASTX727
- 7-Day Schedule (Experimental): 7-Day Schedule
  IMP will be administered for 7 days in total per 4 weeks, i.e. a 28-day cycle.
  Interventions: Drug: ASTX727

INTERVENTIONS:
Drug: ASTX727 — oral decitabine 5mg + cedazuridine
  Arms: 10-Day Schedule
Drug: ASTX727 — oral decitabine 5mg + cedazuridine
  Arms: 5-Day Schedule A
Drug: ASTX727 — oral decitabine 10mg + cedazuridine
  Arms: 5-Day Schedule B
Drug: ASTX727 — oral decitabine 20mg + cedazuridine
  Arms: 5-Day Schedule C
Drug: ASTX727 — oral decitabine 10mg + cedazuridine
  Arms: 7-Day Schedule

SUMMARY:
To investigate the tolerability and safety of ASTX727 in Japanese subjects with lower-risk MDS.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects with a definitive diagnosis of MDS and classified as low or Intermediate-1 risk by the International Prognostic Scoring System (IPSS) risk category
2. Subjects meeting at least one of the disease-related criteria for Red blood cell (RBC) transfusion, hemoglobin (Hb) ,Absolute neutrophil count,Platelet count within 8 weeks prior to initial administration of IMP
3. Subjects with Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
4. Adequate hepatic and renal function
5. Sexually active men with reproductive capacity (except those who have undergone bilateral orchidectomy) must agree to use 2 effective contraceptive measures or remain abstinent during the trial and for 3 months after final administration of IMP. Sexually active women of child-bearing potential must agree to use 2 effective contraceptive measures or remain abstinent during the trial and for 6 months after final administration of IMP.
6. Subjects who have provided written informed consent using the form approved by the institutional review board

Key Exclusion Criteria:

1. Subjects who have received cytokine therapy, immunosuppressant therapy, or chemotherapy within 4 weeks prior to initial investigational medicinal product (IMP) administration
2. Subjects who have received any other IMP or privately-imported medicine within 2 weeks prior to initial IMP administration
3. Subjects with deletion 5q who are to be treated with lenalidomide
4. Subjects with current or previous bone marrow blast percentage of >10%
5. Subjects with a diagnosis of chronic myelomonocytic leukemia
6. Subjects with heart disease of New York Heart Association (NYHA) Functional Class 3 or 4
7. Subjects with an uncontrolled systemic disease or active uncontrolled infection
8. Subjects with diabetes mellitus requiring medical treatment
9. Subjects with a life-threatening illness, medical condition or multiple organ dysfunction, or other reason, including laboratory abnormalities, which in the investigator's or subinvestigator's opinion could compromise the subject's safety, interfere with the absorption or metabolism of IMP, or compromise the integrity of the trial outcome
10. Subjects with prior malignancy
11. Subjects who test positive for human immunodeficiency virus antibody, hepatitis B virus DNA, or hepatitis C virus antibody
12. Subjects with a history of surgical gastrectomy
13. Subjects with previous organ transplantation
14. Subjects with a ≥Grade 2 AE attributable to treatment of underlying disease, excluding the AEs
15. Subjects who have undergone an invasive and extensive operation within 2 weeks prior to initial IMP administration
16. Subjects with hypersensitivity to the IMPs or their excipients
17. Subjects with known significant mental illness or other condition, such as active alcohol or other substance abuse or addiction, that in the opinion of the investigator or subinvestigator predisposes the subject to high risk of noncompliance with the protocol
18. Female subjects who are pregnant, breast-feeding, or who test positive for pregnancy at screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 28days

SECONDARY OUTCOMES:
Area under the curve (AUC) | Pre-dose, 15 min, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h after dosing
  pharmacokinetics parameter
Maximum plasma concentration (Cmax) | Pre-dose, 15 min, 30 min, 60 min, 90 min, 2 h, 3 h, 4 h, 6 h, 8 h, 24 h after dosing
  pharmacokinetics parameter

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- NTT Medical Center Tokyo, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
The focus of this study is a rare disease.